CLINICAL TRIAL: NCT07369843
Title: Effects of Low Power LASER on the Heart Rate Variability of Human Subjects
Brief Title: LASER Effects Blood Flow
Acronym: LASERBF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Paul's Hospital, Congregation Of The Sisters Of Saint Paul De Chartres (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LASERBF1; Saint Paul's Hospital (Other: Saint Paul's Hospital)
Record Dates: First submitted 2025-09-26; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-07

CONDITIONS: Pain Management
Keywords: low power LASER; Heart rate; autonomic tone
MeSH Terms: conditions — Agnosia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test effect (Experimental): Control, experiment, and recovery data will be acquired for each volunteer
  Interventions: Other: physical therapy (low power LASER)

INTERVENTIONS:
Other: physical therapy (low power LASER) — Low power laser with an intensity for pain relieving will be applied to volunteers

SUMMARY:
This study investigate the potential impact of low power laser (LPL), an non-invasive physical therapy, on the cardiovascular system by focusing on its effect on heart rate and autonomic tone.

Study will recruit healthy volunteers and non-invasively monitor their electrocardiogram and digital pulse in response to LPL.

In addition, the potential involvement of autonomic tone will be clarify by topically applying gel (2% lidocaine gel)

DETAILED DESCRIPTION:
This study investigate the potential impact of low power laser (LPL), an non-invasive physical therapy, on the cardiovascular system by focusing on its effect on heart rate and autonomic tone.

Study will recruit healthy volunteers (age 20-60; having no diabetes, hypertension, or other medical problem) and non-invasively monitor their electrocardiogram and digital pulse in response to LPL (with an intensity for relieving pain).

In addition, the potential involvement of autonomic tone will be clarify by topically applying gel (2% lidocaine gel) at the site 2 cm distal to the applying site.

ELIGIBILITY:
Inclusion Criteria:

* age from 20-45

Exclusion Criteria:

* no medical history of diabetes, hypertension, or other medical problem

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
heart rate | Continuous heart rate (HR) recording will start when it is stable after a brief resting (10 min); maintained during stimulation (30 min), and lasted for a period until the HR recovers.
  the heart rate before, during, and after low power LASER